CLINICAL TRIAL: NCT05600933
Title: Prospective Procurement of Tumor Tissue to Identify Novel Therapeutic Targets and Study the Tumor Microenvironment
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000958; 000958-C
Record Dates: First submitted 2022-10-25; First posted 2022-11-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09-09

CONDITIONS: Solid Tumors; Hematologic Malignancy; Gastrointestinal Cancer; Liver Cancer; Pancreatic Cancer; Melanoma; Pre-Malignancy; Lung Cancer
Keywords: Biologic Samples; Intratumoral Immunologic Landscape; Tumor Infiltrating Lymphocytes; Immuno-Oncology Therapeutics; Natural History
MeSH Terms: conditions — Hematologic Neoplasms; Gastrointestinal Neoplasms; Liver Neoplasms; Pancreatic Neoplasms; Melanoma; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 - premalignant, primary or metastatic solid tumor: Participants >= 18 with a suspected or confirmed solid tumor malignancy that requires surgery or biopsy.
- 2 - known or suspected hematologic malignancy: Participants >= 18 who have a known or suspected hematologic malignancy that requires surgery or biopsy.

SUMMARY:
Background:

Many advances have been made in cancer treatments, but more research is needed. Comparing samples of cancerous tissue to samples of normal, noncancerous tissues may help find differences between them. These differences may help researchers find new ways to treat cancer.

Objective:

To collect tissues and blood samples from people with known or suspected cancer. The samples will be used to help identify new targets for cancer treatments.

Eligibility:

People aged 18 years and older with a known or suspected cancer that requires surgery or biopsy.

Design:

Participants will be screened. They will answer questions about their health. They can do this on the phone or in person.

Researchers will collect information from participants medical records. Data may include information about any prior or current cancers. Data about other medical conditions may also be collected.

Participants will have blood drawn. Some of the blood will be tested for HIV and hepatitis B and C. Some of the blood will be used for genetic research.

Participants will have tissue samples collected during surgeries or biopsies. These are procedures the participants would have had as part of their standard care. No new procedures will be done just for this study. Researchers may also seek out samples from prior procedures the participant had done.

Participants will remain in the study for 6 months. They may have blood drawn again. Researchers may also collect tissue samples from any procedures performed during that time.

DETAILED DESCRIPTION:
Background:

* Recent advances and insights into the molecular pathogenesis of cancer have led to the development of novel molecular and biologic targeted therapies for the treatment of advanced cancer participants. A critical challenge in extending these studies involves the identification and validation of new therapeutic targets for future cancer therapies.
* The development of immuno-oncology therapeutics across a wide spectrum of malignancies has emphasized a need to understand the intratumoral immunologic landscape of metastatic cancer. The techniques of cultivating and examining tumor infiltrating lymphocytes developed in the Surgery Branch can be expanded and refined by the exploration of solid tumors.
* The Surgery Branch, NCI has an interest in identifying novel molecular and biologic targets to facilitate the development of future cancer therapies for solid and hematologic malignancies. Through close collaborations with the Surgical Oncology Program and Thoracic Surgery Branch, our internal staff surgeons, and our medical oncology staff clinicians, we are uniquely positioned to acquire and perform important studies on solid tumor tissue and bone marrow to help identify therapeutic targets that may have significant clinical ramifications.

Objective:

To collect biologic samples from participants undergoing diagnostic or therapeutic interventions for known or suspected cancer for the purpose of identifying novel molecular and biologic therapeutic targets and studying the intratumoral immune landscape.

Eligibility:

Participants >=18 years of age with suspected or confirmed malignancies planning diagnostic or therapeutic intervention from which biologic samples may be obtained.

Design:

* A tissue acquisition trial in which tissues will be obtained at the time of intervention.
* Tissue and blood will be processed at the time of collection, stored and then transferred to the Surgery Branch Cell Production Facility for further processing.
* No investigational therapy will be given.
* It is anticipated that 1200 participants will be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age >= 18 years
* Willing to undergo serologic testing for HIV, hepatitis B and C
* Participants who have a known or suspected cancer that requires surgery or biopsy as a part of the standard of care diagnosis, treatment and/or follow up.

Note: Participants will not be enrolled exclusively for the procurement of tissue samples.

-Able and willing to sign an informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from both sexes and all racial/ethnic groups who are undergoing diagnostic or therapeutic interventions for premalignant, primary or metastatic solid tumors or hematologic malignancies
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2033-06-15 (Estimated); Study Completion 2033-06-15 (Estimated)

PRIMARY OUTCOMES:
To collect biologic samples from participants undergoing diagnostic or therapeutic interventions for premalignant, primary or metastatic solid tumors and hematologic malignancies | At time of surgery or biopsy
  To collect biologic samples from participants undergoing diagnostic or therapeutic interventions for known or suspected cancer for the purpose of identifying novel molecular and biologic therapeutic targets and studying the intratumoral immune landscape.

SECONDARY OUTCOMES:
To collect detailed history, demographic, treatment data, and perioperative findings. | At time of consent
  To collect detailed history, demographic, treatment data, and perioperative findings in order to categorize specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.@@@@@@Genomic data will be available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data will be made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000958-C.html